CLINICAL TRIAL: NCT01352143
Title: Measurements of Thrombin Generation in Response to Recombinant Activated Factor VII and Prothrombin Complex Concentrate in Neonatal Plasma After Cardiopulmonary Bypass
Brief Title: Thrombin Generation in Neonatal Plasma After Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's Research Oversight Committee Funds (Unknown)
Responsible Party: Principal Investigator, Nina Guzzetta, M.D., Associate Professor of Anesthesiology, Emory University
Other Study IDs: IRB00048151
Record Dates: First submitted 2011-04-20; First posted 2011-05-11 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Cardiopulmonary Bypass
Keywords: Neonates
MeSH Terms: interventions — Factor IX; factor IX, factor VII, factor X, prothrombin drug combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples only
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Recombinant activated factor VII — Plasma will be spiked in vitro with recombinant activated factor VII to assess increases in thrombin generation with and without the drug
  Other Names: NovoSeven RT, Novo Nordisk, Bagsvaerd, Denmark
Drug: Prothrombin Complex Concentrate — Plasma will be spiked in vitro with prothrombin complex concentrate to determine increases in thrombin generation with and without the drug
  Other Names: Beriplex P/N, CSL Behring, King of Prussia, PA

SUMMARY:
The primary goal of this investigation is to determine the ability of recombinant activated factor VII (rFVIIa) and prothrombin complex concentrate (PCC) to improve thrombin generation in neonatal plasma after CPB.

DETAILED DESCRIPTION:
In this investigation, the investigators propose a comparison in vitro of the ability of rFVIIa with that of PCC to increase thrombin generation in neonatal plasma after CPB. A pre-cardiopulmonary bypass (CPB) baseline blood sample will be obtained. After the termination of CPB and the administration of one round of protamine, platelets and fibrinogen (standard of care), a second blood sample will be drawn. All samples will be centrifuged to yield platelet rich plasma and stored until processing. In the pre-CPB sample, baseline thrombin generation will be measured. The post-CPB sample will be divided into three aliquots to measure thrombin generation under three different circumstances: the first will serve as a control, the second will include rFVIIa and the third PCC.

ELIGIBILITY:
Inclusion Criteria:

1. Full-term neonates (36-42 weeks gestational age)
2. Apgar score of 7 or more at 5 minutes after delivery
3. Neonates undergoing elective cardiac surgery requiring CPB at Children's Healthcare of Atlanta at Egleston
4. Parents willing to participate, and able to understand and sign the provided informed consent

Exclusion criteria:

1. Preterm neonates (less than 36 weeks gestation)
2. Apgar score of less than 6 at 5 minutes after birth
3. Emergent procedure
4. Patients undergoing cardiac surgery not requiring CPB
5. Neonates with a known coagulation defect or coagulopathy
6. Mother with a known coagulation defect or coagulopathy
7. Parents unwilling to participate or unable to understand and sign the provided informed consent

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates (less than 30 days of age) undergoing complex congenital cardiac surgery requiring cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Peak thrombin Generation | one year
  The primary outcome measure is the peak amount of thrombin generated (measured in nM) as determined by the Thrombinoscope with rFVIIa as compared to PCC.

CONTACTS AND LOCATIONS:
Overall Officials: Nina A Guzzetta, M.D., Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States